CLINICAL TRIAL: NCT03557060
Title: NUCALA ® Subcutaneous Injection Special Drug Use Investigation (EGPA, Long-term）
Brief Title: NUCALA® Special Drug Use Investigation (EGPA, Long-term)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208505
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Churg-Strauss Syndrome; Eosinophilic Granulomatosis With Polyangiitis
Keywords: Nucala; Drug use investigation; EGPA; Long-term
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects receiving NUCALA: Subjects with a diagnosis of EPGA, for which NUCALA is indicated will be included.
  Interventions: Drug: Nucala

INTERVENTIONS:
Drug: Nucala — NUCALA injections will be administered to eligible subjects with diagnosis of EGPA. Dose unit, daily dose frequency, date of administration will be at the investigator discretion.

SUMMARY:
This study is a drug use investigation program of NUCALA. The objective of this study is to collect and assess information on the safety and effectiveness of the long-term use of NUCALA SC injection in daily clinical practice in subjects with Eosinophilic Granulomatosis with Polyangiitis (EGPA). All subjects who administered NUCALA for the treatment of EGPA after its approval of indication will be included in the study. In addition, after the approval, subjects who had already received NUCALA for EGPA prior to the conclusion of the contract will also be included. Approximately 300 subjects will be included in the study. The observation period per subject is up to 96 weeks (2 years) from the start of NUCALA administration for EGPA at a maximum. If a subject has withdrawn from/terminated administration of NUCALA, it will be until the withdrawal/termination. Additionally, to consider the safety and effectiveness of NUCALA administration in subjects who had withdrawn from/terminated due to symptom improvement, 48 weeks (1 year) follow-up investigation should be conducted as much as possible. The total study duration will be approximately 3 years (2 years observation period and 1 year follow-up) from the approval of EGPA indication to the lifting of approval condition. NUCALA is a registered trademark of the GlaxoSmithKline [GSK] group of companies.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who administered NUCALA for the treatment of EGPA after its approval of indication will be included in the study. In addition, after the approval, subjects who had already received NUCALA for EGPA prior to the conclusion of the contract will also be included.
* Subjects who had been registered to NCT03028480 for bronchial asthma, but had a change in treatment purpose from bronchial asthma to EGPA during the observation period

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who administered NUCALA for the treatment of EGPA after its approval of indication will be included in the study.
Sampling Method: Probability Sample
Enrollment: 4115 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions | Up to 2 years
  The information regarding the incidences of adverse drug reactions will be collected.
Response rate based on global assessment of effectiveness | Up to 2 years
  The response rate is the percentage of subjects assessed as effective. Effectiveness will be comprehensively assessed by any of effective or not effective at Week 12, 48 after the start of NUCALA administration, end of the observation period, or withdrawal/termination, based on the course of subjective symptoms, course of clinical symptoms, from the start date of administration to the end of the observation period. If effectiveness cannot be determined for some reasons, it should be assessed as indeterminable and its reasons should be recorded on the CRF.
Time to EGPA remission and recurrence | Up to 2 years
  The time to EGPA remission and recurrence will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan

REFERENCES:
- [Background] Fujii T, Atsumi T, Okamoto N, Takahashi N, Tamura N, Nakajima A, Nakajima A, Matsuno H, Mukai I, Ishida A, Aizawa K, Kuwana M, Takagi M, Takeuchi T.Post-marketing surveillance of mepolizumab use in patients with eosinophilic granulomatosis with polyangiitis in Japan: Interim analysis.Ther Res.2021;42(6):403-422